CLINICAL TRIAL: NCT06769776
Title: Drain Versus No-Drain After Live Donor Hepatectomy- A Randomized Controlled, Pilot Study
Brief Title: Drain vs No Drain After Live Donor Hepatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marengo Asia Hospitals (Other)
Responsible Party: Principal Investigator, Bharat Nair, Principle Investigator. Consultant , Department of HPB surgery and liver Transplant, Marengo Asia Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MAHF/AP/LTP-1/EC/2024/04
Record Dates: First submitted 2024-08-05; First posted 2025-01-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Donor Hepatectomy

STUDY DESIGN:
Intervention Model Description: The investigators aim to compare the safety of no drain placement vs abdominal drain placement in LDLT by comparing the comprehensive complication index(CCI) between both arms at day of discharge after donor hepatectomy.
Masking Description: Trial will commence as soon as clearance from ethics committee is achieved. All voluntary healthy liver donors planned for donor hepatectomy, fulfilling inclusion criteria and not matching any of the exclusion criteria will be recruited . On the day of surgery, donor will be alloted either of the arms based on computer generated block randomization code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain (No Intervention): Patients in the drain arm will undergo routine steps in donor hepatectomy. After graft removal, hemostasis and biliostasis will be confirmed, following which at the end of the operation ,a 28 Fr abdominal drain will be inserted with tip near cut surface of remnant
- No Drain (Experimental): Patients in the no drain arm will undergo routine steps in donor hepatectomy. After graft removal, hemostasis and biliostasis will be confirmed, following which abdomen will be closed in layers. No intraabdominal drain will be placed.
  Interventions: Other: No Drain i.e. Omission of abdominal drain placement

INTERVENTIONS:
Other: No Drain i.e. Omission of abdominal drain placement — Omission of abdominal drain placement in intervention arm. The No-drain arm will be compared to drain arm
  Arms: No Drain

SUMMARY:
Prophylactic abdominal drain placement after donor hepatectomy has been a common or even mandatory practice in most transplant centers. This serves to monitor the occurrence of post-operative intra-abdominal bleeding and is used for the detection and drainage of any bile leakage. However prophylactic drain placement is not without complications, like; Increased rates of intraabdominal and wound infection, Increased abdominal pain, Decreased pulmonary function, Bowel injury and Prolonged hospital stay. Comprehensive Complication Index (CCI) is a valuable tool used to assess the overall morbidity of patients after surgical interventions . The CCI score ranges from 0 (no complication) to 100 (death), reflecting the gravity of the overall complication burden on the patient on a continuous scale and is a validated tool for living donor liver transplants. The investigators aim to compare the safety of no drain placement vs abdominal drain placement in LDLT(Live Donor Liver Transplant) by comparing the comprehensive complication index(CCI) between both arms at day of discharge after donor hepatectomy.

DETAILED DESCRIPTION:
* This study will be a randomised controlled, pilot study to compare the safety of no drain placement vs abdominal drain placement in LDLT by comparing the comprehensive complication index(CCI) between both arms at day of discharge after donor hepatectomy.
* Patient admitted for donor hepatectomy will be recruited and further randomised into the Drain and No-Drain arms. Patients in the no drain arm will undergo routine steps in donor hepatectomy. After graft removal, hemostasis and biliostasis will be confirmed, following which abdomen will be closed in layers. For patients in the drain arm, same steps will be followed. At the end of the operation , additionally, 28 Fr abdominal drain will be inserted with tip near cut surface of remnant. Intraoperative and post-operative parameters will be compared between the groups. Comprehensive Complication index will be calculated on day of discharge using online universal CCI calculator application.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing donor hepatectomy -

Exclusion Criteria:

Any patient not consenting to the procedure. Intraoperative need for drain placement in no drain arm due to surgical factors.

Inverted L/ J shaped incision. Laparoscopic donor hepatectomy Robotic donor hepatectomy.

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
CCI index on post operative day 7 | Admission one day prior to live donor hepatectomy till post operative day 7.
  Comprehensive Complication Index (CCI) is a valuable tool used to assess the overall morbidity of patients after surgical interventions . The CCI score ranges from 0 (no complication) to 100 (death), reflecting the gravity of the overall complication burden on the patient on a continuous scale and is a validated tool for living donor liver transplants. The investigators aim to compare the safety of no drain placement vs abdominal drain placement in LDLT by comparing the comprehensive complication index(CCI) between both arms on post operative day 7 after donor hepatectomy.

SECONDARY OUTCOMES:
Infective complications | Admission one day prior to live donor hepatectomy till post operative day 7
  Surgical site infections, intra abdominal abscesses
Duration of hospital stay | Admission one day prior to live donor hepatectomy till post operative day 7
  Total days of hospitalization required from admission till post operative day 7
Paralytic ileus | Admission one day prior to live donor hepatectomy till post operative day 7.
  Days to start normal oral diet after surgery
Bile leak | Admission one day prior to live donor hepatectomy till post operative day 7
  Occurrence and detection of bile leak after donor hepatectomy
Hemorrhage | Admission one day prior to live donor hepatectomy till post operative day 7
  Occurrence and detection of bleeding after live donor hepatectomy
Post operative pain scores | Admission one day prior to live donor hepatectomy till post operative day 7
  Post operative pain as measured by twice daily (Visual Analogue Scale)VAS scores

CONTACTS AND LOCATIONS:
Overall Officials: Punit Singla, MS,DNB, Study Director — Marengo Asia Hospitals
Locations (1):
- Marengo Asia Hospitals, Faridabad, Haryana, India

IPD SHARING:
Plan to Share IPD: No
Name or address in the study data will be coded with initials and number . The confidentiality will be maintained. Unless required by law, only the Study Doctor, the Study Team and its authorized agents and the Ethics Committee/Institution Review Board will have access to confidential data which identifies patients by name or has access to the in patient records of the patient